CLINICAL TRIAL: NCT05785754
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Expansion Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of DCSZ11 as a Monotherapy and in Combination in Patients With Advanced or Metastatic Solid Tumors
Brief Title: DCSZ11 as a Monotherapy and in Combination in Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: DynamiCure Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCSZ11-101
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab; Doxorubicin; tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1a Dose Escalation Monotherapy (Experimental): Dose escalation to investigate the safety and tolerability of DCSZ11.
  Interventions: Drug: DCSZ11
- Phase 1a Dose Escalation Combination (Experimental): Dose escalation to investigate safety and tolerability, and determine DCSZ11 Phase 1b doses in combination with pembrolizumab.
  Interventions: Drug: DCSZ11; Drug: Pembrolizumab
- Phase 1b Dose Expansions (Experimental): Dose expansion to further investigate the safety, tolerability, and preliminary evidence of antitumor activity of the combination with pembrolizumab in select tumor indications.
  Interventions: Drug: DCSZ11; Drug: Pembrolizumab
- Phase 1b Standard of Care (Experimental): Phase 1b - Standard-of-Care (SOC) Combinations Safety Lead-in/ Expansion in Select Indications A safety lead-in using the BOIN design followed by a Simon two-stage like design will be used to evaluate DCSZ11 in combination with standard of care in select indications. Patients will receive DCSZ11 IV at one of the dose escalation dose levels/schedule (or dose/schedule selected for optimization/expansion). Once the safety lead-in is completed, a Bayesian continuous toxicity monitoring will be used to monitor for unacceptable toxicity in expansions.
  The following SOC combination expansion cohorts will be enrolled:
  * 1b SOC Cohort 1: Doxorubicin combination in soft tissue sarcoma
  * 1b SOC Cohort 2: Tebentafusp combination in uveal melanoma
  Interventions: Drug: Doxorubicin; Drug: Tebentafusp

INTERVENTIONS:
Drug: DCSZ11 — A monoclonal antibody that binds to CD93, DCSZ11 will be administered as a single intravenous (IV) infusion on Day 1 in each 21-day cycle.
  Arms: Phase 1a Dose Escalation Combination; Phase 1a Dose Escalation Monotherapy; Phase 1b Dose Expansions
Drug: Pembrolizumab — Pembrolizumab injection
  Arms: Phase 1a Dose Escalation Combination; Phase 1b Dose Expansions
Drug: Doxorubicin — 1b SOC Cohort 1: Doxorubicin combination in soft tissue sarcoma
  Arms: Phase 1b Standard of Care
Drug: Tebentafusp — 1b SOC Cohort 2: Tebentafusp combination in uveal melanoma
  Arms: Phase 1b Standard of Care

SUMMARY:
This is a multicenter, open-label, Phase 1 study to assess the effects of DCSZ11 as a monotherapy and in combination in patients with advanced or metastatic solid tumors. The study consists of an Escalation Phase (Phase 1a) and a Dose Expansion/Optimization Phase (Phase 1b).

DETAILED DESCRIPTION:
DCSZ11 will be administered as monotherapy and in combination with pembrolizumab in patients with advanced-stage or metastatic solid tumors. The Escalation Phase will be followed by a Dose Expansion/Optimization Phase (Phase 1b) to further characterize safety, PK, pharmacodynamics, and evidence of antitumor activity of DCSZ11 in combination with pembrolizumab in select relapsed/refractory (R/R) solid tumors and, if desired, optimize the DCSZ11 dose.

Phase 1a - Dose Escalation Phase 1a is a dose escalation study of DCSZ11 as monotherapy in Part 1 and in combination with pembrolizumab in Part 2. DCSZ11 dose levels may be escalated up to the maximum tolerated dose level or to the maximum planned dose level of 20mg/kg. Patients will receive DCSZ11 IV initially every 3 weeks.

Phase 1b - Dose Expansion/Optimization in Select Indications Phase 1b will evaluate DCSZ11 in combination with pembrolizumab in select indications following a Simon two-stage like design that allows for dose optimization.

Phase 1b - Standard-of-Care (SOC) Combinations Safety Lead-in/ Expansion in Select Indications A safety lead-in using the BOIN design followed by a Simon two-stage like design will be used to evaluate DCSZ11 in combination with standard of care in select indications. Patients will receive DCSZ11 IV at one of the dose escalation dose levels/schedule (or dose/schedule selected for optimization/expansion). Once the safety lead-in is completed, a Bayesian continuous toxicity monitoring will be used to monitor for unacceptable toxicity in expansions.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Be willing and able to provide written informed consent for the study.
3. Patients in Phase 1a must have a histologically or cytologically documented, advanced (metastatic and/or unresectable) solid tumor that has progressed on or after standard therapy (relapsed/refractory patients; patients must have failed at least one prior line of therapy) or for whom there is no effective standard therapy based on the Investigator's judgment.

   Note: Patients with glioblastoma (GBM) or other central nervous system(CNS) tumors may participate if they are on stable or decreasing corticosteroid levels not exceeding 2 mg/day dexamethasone (or equivalent doses of other corticosteroids) within 7 days of the first dose of study drug or do not require corticosteroids.

   Note: For patients who are intolerant to or refuse standard-of-care therapy for recurrent disease, reasons must be documented.
4. Patients in Phase 1b Dose Optimization/Expansion must have one of the following:

   1. Non-squamous NSCLC for which prior standard first-line treatment containing an anti-PD-(1/L1) checkpoint inhibitor alone or in combination has failed and that has progressed to no more than 2 prior systemic therapies. Patients must not have presented with disease progression during the first 3 months of treatment with first line anti-PD-(1/L1)-containing therapy. Patients must have had documented disease progression per RECIST 1.1 within 12 weeks from the last dose of anti-PD-1/L1 mAb to be considered to have failed an anti-PD-(1/L1) mAb containing therapy. The initial evidence of disease progression to anti-PD-1/L1 mAb containing therapy needs to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression.

      Note: Patients with known driver mutations/genomic aberrations (i.e., EGFR, B-Raf proto-oncogene mutation V600E [BRAF V600E], and ROS proto-oncogene 1 [ROS1] sensitizing mutations, neurotrophic receptor tyrosine kinase [NRTK] gene fusions, and ALK rearrangements) are not eligible.

      Note: Patients with rapid clinical progression are excluded from participation.
   2. Immunotherapy-naïve microsatellite stable-CRC (MSS-CRC) that failed or was intolerant to ≥ 2 lines of therapy and that progressed on/after no more than 4 lines of therapy.

   Note: Patients must have received prior treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-containing regimens if indicated. Patients eligible for treatment with an approved and available targeted therapy must have been offered such therapy prior to enrollment. Adjuvant chemotherapy will be considered a prior line of therapy if the patient progressed while on or within 6 months of completing adjuvant treatment.
5. Patients in Phase 1b Standard-of-Care Combination Lead-in/Expansions must have one of the following:

   1. Histologically confirmed, anthracycline naïve, metastatic or locally advanced, unresectable soft-tissue sarcoma for which doxorubicin monotherapy is indicated. Note: Ewing sarcoma, gastrointestinal stromal tumor (GIST), and Kaposi sarcoma are excluded.
   2. Histologically confirmed, metastatic or advanced, unresectable uveal melanoma that are eligible for treatment with tebentafusp monotherapy. Patients should not have received more than 4 doses of tebentafusp at the target dose level of 68 mcg.
6. Patients must have a lesion not previously irradiated that can be biopsied with acceptable clinical risk and agree to have a fresh biopsy at Screening and on treatment; except patients with GBM or other CNS tumors. Every effort must be made to take the second biopsy from the same lesion of the biopsy at Screening.
7. Patients must have at least 1 measurable lesion according to RECIST 1.1; except for patients enrolled in monotherapy dose levels 1 and 2.

   1. A lesion in a previously irradiated area is eligible to be considered as a measurable disease as long as there is objective evidence of progression of the lesion before study enrollment.
   2. Patients must have at least 1 measurable lesion for inclusion that will not undergo biopsy.
   3. Patients with GBM must meet the RANO criteria of measurable disease for the post-gadolinium primary T1WI.
8. Patients with previously treated CNS metastases may participate provided that:

   1. They are stable (i.e., without evidence of progression by magnetic resonance imaging [MRI]) for ≥ 4 weeks prior to the first dose of study drug), and
   2. All neurologic symptoms have returned to baseline, and
   3. For patients enrolled in expansion cohorts, have not required steroid treatment for at least 14 days before the first dose of study intervention Patients with signs or symptoms suggestive of CNS metastases, must have brain imaging performed to confirm the absence of detectable CNS disease within 2 weeks prior to the first dose of study drug.

   Note: This criterion does not apply to patients with GBM or other CNS tumors.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. Patients enrolled in expansion cohorts must have an ECOG performance status of 0 or 1.
10. Adequate organ function and bone marrow reserve as indicated by the following laboratory assessments performed within 10 days prior to the first dose of study drug:

    1. Bone marrow function: absolute neutrophil count (ANC) ≥ 1000/µL, ANC ≥ 1500/µL in expansions; hemoglobin ≥ 9 g/dL (criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks) ; platelet count ≥ 75,000/µL, platelet count ≥ 100,000/µL in expansions.
    2. Hepatic function: Total serum bilirubin ≤ 1.5 × the upper limit of normal (ULN) or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN; serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT), ≤ 2.5 × ULN (≤ 5 × ULN in the presence of hepatic metastases).

       Note: Patients with inherited disorders of bilirubin metabolism should be discussed with the Sponsor.
    3. Renal function: Creatinine clearance ≥ 30 mL/minute based on Cockcroft-Gault estimation.
    4. Coagulation profile: Prothrombin time (PT)-international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Patients on a stable, maintenance regimen of anticoagulant therapy for at least 30 days prior to the first dose of study drug may have PT/INR measurements > 1.5 × ULN if, in the opinion of the Investigator, the patient is suitable for the study. An adequate rationale must be provided to the Sponsor prior to enrollment.
11. Have recovered to Grade 1 or baseline from all toxicity associated with previous therapy or have the toxicity established as sequela.

    Note: Neuropathy and/or hearing impairment ≤Grade 2, any grade alopecia, or autoimmune endocrinopathies with stable replacement therapy are permitted.
12. Patients receiving a combination with standard-of-care must meet established treatment criteria for the respective standard-of-care agent(s).
13. Patients with human immunodeficiency virus (HIV) must have well controlled disease on antiretroviral therapy (ART), defined as:

    1. Patients on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening.
    2. Patients on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening.
    3. Patients on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study.
    4. Patients must not have had any AIDS-defining opportunistic infections within the past 12 months or any history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
14. Female patients must agree to not breastfeed through 5 months after the last dose of study drug and must meet 1 of the following:

    1. Postmenopausal for at least 1 year before the screening visit, or
    2. Surgically sterile, or
    3. Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing of the ICF through 5 months after the last dose of study, or
    4. Agree to practice true abstinence during the entire study treatment period and through 5 months after the last dose of study drug, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.
15. Male patients, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following:

    1. Agree to practice effective barrier contraception from the time of signing of the ICF through 2 months after the last dose of DCSZ11, or
    2. Agree to practice true abstinence from the time of signing of the ICF through 2 months after the last dose of study drug, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.
16. Must be willing and able to comply with clinic visits and procedures outlined in the study protocol.

Criteria for Exclusion:

1. Received systemic anticancer treatments or investigational products within 28 days before the first dose of study drug or 5 half-lives, whichever is shorter.

   Note: Low-dose steroids (oral prednisone ≤10 mg per day or equivalent), hormonal therapy for prostate cancer or breast cancer (as adjuvant treatment), and treatment with bisphosphonates and receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitors are allowed.
2. Received extended field radiotherapy ≤4 weeks before the start of treatment (≤7 days for limited field radiation for palliation outside the chest or brain) or has radiation related toxicities requiring corticosteroid treatment.
3. Patients with second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the patient is not on active anticancer therapy. These patients must be discussed with the Sponsor prior to enrollment.
4. Patients with known active CNS metastases and or carcinomatous meningitis.
5. Systemic arterial thrombotic or embolic events, such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 3 months prior to the first dose of study drug
6. Systemic venous thrombotic events (e.g., deep vein thrombosis) or pulmonary arterial events (e.g., pulmonary embolism) within 1 month prior to the first dose of study drug. Patients with venous thrombotic events prior to the first dose of study drug on stable anticoagulation therapy are eligible.
7. Left ventricular ejection fraction (LVEF) < 50%.
8. Major surgery within 4 weeks and minor surgery within 2 weeks of the first dose of study drug; following surgeries, all surgical wounds must be healed and free of infection or dehiscence. Patients must have recovered and not have ongoing surgical complications.
9. Marked proteinuria ≥ 2 g/24 hours and/or nephrotic syndrome. Patients with proteinuria 2+ or greater urine dipstick reading should undergo further assessment, e.g., a 24-hour urine collection.
10. Known allergy or hypersensitivity to any component of the study drugs or, for patients receiving the imaging agent, any component of the imaging agent.
11. For patients receiving a combination with pembrolizumab:

    1. Received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
    2. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
    3. Autoimmune disease requiring systemic immunosuppressive therapy within the past 2 years. Hormone therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered an excluded form of systemic treatment of an autoimmune disease.
    4. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
    5. History of radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study treatment
    6. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
    7. History of allogeneic tissue or solid organ transplant.
12. Receipt of any live or live-attenuated vaccine within 4 weeks of initiation of study treatment. Administration of killed vaccines is allowed.
13. Has active infection requiring systemic therapy.
14. Patients that are hepatitis B virus surface antigen (HBsAg) seropositive and with detectable hepatitis B virus (HBV) viral load. Note: Patients with positive HBsAg can been enrolled if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to initiation of study treatment. Patients should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.
15. Patients with history of hepatitis C virus (HCV) infection and detectable HCV viral load at screening. Note: Patients must have completed curative antiviral therapy at least 4 weeks prior to initiation of study treatment.
16. History of any of the following ≤6 months before first dose: congestive heart failure New York Heart Association Grade III or IV, unstable angina, myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, ongoing symptomatic cardiac arrhythmias >Grade 2, or any other serious cardiac condition (e.g., pericardial effusion or restrictive cardiomyopathy). Chronic atrial fibrillation on stable anticoagulant therapy is allowed.
17. History or current evidence of any condition, therapy, laboratory abnormality, psychiatric illness, social circumstances, or other circumstance that might compromise the ability to provide informed consent, confound the results of the study, or interfere with the patient's ability to cooperate with the requirements of the study, such that it is not in the best interest of the patient to participate, in the opinion of the treating investigator.
18. Female patients who are pregnant or lactating and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Incidence of dose limiting toxicites (DLTs) | 21 days
Phase 1a: Frequency and severity of treatment emergent adverse events | up to 3 years
Phase 1b: Overall response rate (ORR) per Investigator-assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST) | 1 year

SECONDARY OUTCOMES:
Phase 1a: Overall response rate (ORR) per Investigator-assessed RECIST v1.1 | 1 year
Phase 1a and b: Overall response rate (ORR) per Investigator-assessed consensus guideline developed by the RECIST Working Group for the use of modified RECIST, Version 1.1 in cancer immunotherapy trials (iRECIST) | 1 year
Phase 1a and b: Duration of response (DOR) as determined per Investigator assessment by RECIST v1.1 and iRECIST | 1 year
Phase 1 a and b: Disease control rate (DCR) as determined per Investigator assessment by RECIST v1.1 and iRECIST. | 1 year
Phase 1a and b: Progression free survival (PFS) as determined per Investigator assessment by RECIST v1.1 and iRECIST. | 3 years
Phase 1 a and b: Overall survival (OS) | 3 years
Phase 1 and b: Pharmacokinetic parameters of DCSZ11 | 2 years
Phase 1 a and b: Incidence of anti-drug antibody (ADA) and neutralizing antibodies (NAbs) against DCSZ11 | 2 years

CONTACTS AND LOCATIONS:
Locations (35):
- United States (14):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute Denver Healthone, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - MonteFiore, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
- Australia (12):
  - Scientia Clinical Research, Randwick, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - University of Sunshine Coast, Buderim, Queensland
  - Southern Oncology Clinical Research Unit (SOCRU), Bedford Park, South Australia
  - The Queen Elizabeth Hospital (TQEH), Woodville South, South Australia
  - Monash Health, Clayton, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
  - Townsville Hospital, Douglas
  - Liverpool Hospital, Liverpool
  - Mater Misericordiae Health Services Brisbane Ltd, South Brisbane
  - Sydney Adventist Hospital, Wahroonga
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-a University Hospital, Busan
  - Cha University Bundang Medical Center, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No